CLINICAL TRIAL: NCT05901792
Title: The Effect of Virtual Reality Games on Changing the Center of Gravity Location in Children With Adolescent Idiopathic Scoliosis
Brief Title: Effect of VRGs on Changing the Center of Gravity Location in AIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assistant professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: E-74555795-050.01.04-689324
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Body statics; spine; rehabilitation technology; Posture; Virtual Reality Games; Center of gravity; Active video games; Scoliosis; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Games (Experimental): VRGs group will receive games that focus on changing the position of the body center of gravity and improving balance levels.
  Interventions: Other: Virtual Reality Games
- Control group (Other): As the control group, the cases on the waiting list will be evaluated.
  Interventions: Other: Waiting List

INTERVENTIONS:
Other: Virtual Reality Games — Six different Nintendo Wii Fit Plus games will be employed for six weeks, three days a week, for a total of 18 sessions ranging from 40 to 60 minutes. The games will be chosen from those that emphasize shifting the body's center of gravity. In addition, participants will be given basic correction exercises (derotation, deflexion, basic tension, and lateral flexion 3*3) at the beginning of the study and instructed to practice them at home for six weeks.
  Arms: Virtual Reality Games
Other: Waiting List — As the control group, the cases on the waiting list will be evaluated. The control group will be given basic elements of corrective exercises (derotation, deflexion, basic tension, and lateral flexion 3*3) at the start of the study and instructed to practice at home for six weeks.
  Arms: Control group

SUMMARY:
The purpose of this clinical trial is to examine the effect of virtual reality games (VRG) on changing the location of the center of gravity in children with adolescent idiopathic scoliosis (AIS).

Twenty-four patients with AIS will be randomly allocated to two groups. The intervention group will apply to the virtual reality games and basic correction exercises group for six weeks (18 sessions). The control group will be given the basic correction exercises. Patients' center of gravity (Physiosoft Balance System), posture parameters (PostureScreen Mobile, Posterior Trunk Asymmetry Index (POTSI) and Anterior Trunk Asymmetry Index (ATSI)), cosmetic perception (Walter Reed Visual Evaluation Scale (WRVAS)) will assess at the first session and the end of 6 weeks.

DETAILED DESCRIPTION:
The most common type of scoliosis is adolescent idiopathic Scoliosis (AIS). It affects 1-4% of adolescents. AIS is associated with cosmetic problems, pain, functional limitations, respiratory dysfunction and a decrease in quality of life. Although scoliosis is characterized by lateral spinal deviation, it causes a three-dimensional deformity with geometric and morphological changes in the trunk and rib cage. The main changes are postural changes in the orientation of the head, shoulders, scapula and pelvis in all three planes, but more specifically rotations of body segments in the horizontal plane. Spinal deformity not only changes the shape of the trunk, but also the relationships between body segments. Therefore, it leads to an abnormal change in the center of gravity. While various treatment approaches are recommended in the management of AIS to overcome these and other complications, scoliosis-specific corrective exercises are almost always part of the treatment plan for individuals with AIS. However ,Virtual Reality Games (VRGs) have recently been used in health and rehabilitation research due to recent technological developments and changes. In the literature, VRGs have been shown to have a positive effect on changing the position of the center of gravity in different rehabilitation areas. However, there is no study examining the effect of the use of VRGs on the chaning of the center of gravity Location in the treatment of AIS.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Adolescent Idiopathic Scoliosis
* Being the Cobb angle between 10 and 25 degrees on the anteroposterior radiograph
* Being between the ages of 11 and 18
* Volunteering to participate in the study

Exclusion Criteria:

* Having a history of spinal surgery and/or tumors
* Using braces and insoles
* Having a positive result of sharpened Romberg and Unterberger test
* Having orthopedic problems affecting the lower extremities that may affect balance
* Having problems with vision and/or hearing
* Having a communication disability
* Having difficulty with understanding given commands
* Having neurological or cognitive impairments
* Receiving conservative treatment for AIS

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Center of gravity | { 6 weeks}
  The physiosoft Balance System is used to assess the location of the body's center of gravity using the Nintendo Wii Fit balance board. This system was developed by engineers and physiotherapists to measure static balance. The physiosoft Balance System is based on the principle of utilizing the Nintendo Wii Fit system through a computer and developing software specifically designed for objective assessment of balance on a balance board. This system evaluated the static standing balance, center of gravity location and postural oscillations of the participants.

SECONDARY OUTCOMES:
Frontal-sagittal plan posture evaluation | { 6 weeks}
  "PostureScreen Mobile" Application: Frontal and sagittal plan posture evaluation will be calculated by marking the reference points on the anterior, posterior and lateral photographs of the patient in "PostureScreen Mobile" application. The total displacement values in the anterior, posterior and lateral directions for postural impairment will be noted in "cm". Decreasing the total displacement values is considered as an improvement in postural parameters.
Body Symmetry-Posterior | { 6 weeks}
  Posterior Trunk Asymmetry Index (POTSI): The Posterior Trunk Asymmetry Index parameter is defined as the sum of the six indices: the three frontal plane asymmetry index (C7, axilla folds and waist lines) and the three frontal plane height difference index (acromions, axilla folds and waist lines). The Posterior Trunk Asymmetry Index score is calculated by placing the indices on the posterior photo of the patient. The Posterior Trunk Asymmetry Index score, which represents full symmetry, is '0' and the increase in score indicates increased trunk asymmetry.
Body Symmetry-Anterior | { 6 weeks}
  Anterior Trunk Asymmetry Index (ATSI): It is defined as the sum of the six indices determined on the patient's anterior photo: three frontal plane asymmetry indices (stern notch, axilla folds and waist lines) and three frontal plane plane height difference indices (acromions, axilla folds and waist lines). The Anterior Trunk Asymmetry Index score is calculated by placing the indices in the formula. The Anterior Trunk Asymmetry Index score, which represents full symmetry, is '0' and the increase in score indicates increased trunk asymmetry.
Deformity perception assessment | { 6 weeks}
  The Walter Reed Visual Assessment Scale (WRVAS): It is designed to understand the visual change caused by scoliosis and evaluates deformity under 7 headings. There are 5 different pictures that show different degrees of deformity. Each deformity is scored from 1 to 5; "1" is the best, "5" is the worst. The total score is obtained by summing the scores from all titles and dividing them by 7. The score ranges from 1 to 5, and a higher total score means that the perceived deformity is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Zengin Alpozgen, Asst. Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)